CLINICAL TRIAL: NCT05559372
Title: Effects of Energy Drink Consumption on Physiological Performance, Mood, and Cardiovascular Outcomes
Brief Title: Energy Drink Effects on Performance, Mood, and Cardiovascular Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nathaniel Jenkins (Other)
Responsible Party: Sponsor-Investigator, Nathaniel Jenkins, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 202107364
Record Dates: First submitted 2022-09-21; First posted 2022-09-29 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Caffeine; Exercise Performance; Energy Drink; Cardiovascular Safety; Mood

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nutrabolt C4 Energy Drink Carbonated (Experimental): 16 oz
  Interventions: Dietary Supplement: Acute energy drink or placebo consumption
- Monster Energy Original (Active Comparator): 16 oz
  Interventions: Dietary Supplement: Acute energy drink or placebo consumption
- Placebo (Placebo Comparator): 16 oz carbonated placebo
  Interventions: Dietary Supplement: Acute energy drink or placebo consumption

INTERVENTIONS:
Dietary Supplement: Acute energy drink or placebo consumption — Participants consumed either 16 oz of Nutrabolt C4 Energy Carbonated, Monster Energy Original, or Placebo in randomized order in three separate visits separated by 7±3 days.

SUMMARY:
Energy drinks are widely promoted to increase energy, enhance mental alertness, and improve physical performance. ccording to the National Center for Complementary and Integrative Health (NCCIH) at NIH [1], next to multivitamins, energy drinks are the most popular dietary supplement consumed by American teens and young adults. No two energy drinks are the same, with each using different ingredients. Traditionally, energy drinks contained caffeine, sugar, ginseng and B-vitamins, but newer competitors are bringing different formulations to the market that are also low-calorie/low-sugar and that contain other performance enhancing ingredients, such as beta-alanine and l-citrulline. There are also significant concerns regarding the safety of energy drink consumption. Unfortunately, there are few studies that have (1) examined the effects of energy drink consumption on performance and cardiovascular safety, nor (2) compared these effects among brands with different formulations to examine their safety and efficacy relative to each other and such studies are desperately needed, especially with the growing popularity of energy drinks [3,4].

DETAILED DESCRIPTION:
After enrollment, subjects will participate in a familiarization visit, followed by 3 separate experimental visits. All of these visits will be separated by ~1 week, and they will occur at approximately the same time of day (±90 minutes). During the familiarization visit, subjects will complete a heath history questionnaire, and then complete brief versions of the study procedures and will be provided with an opportunity to ask questions to ensure that they are comfortable with the tests before beginning the experimental visits. In this study subjects will consume various test beverages that may enhance physiologic performance and mood. Subjects will consume one of these beverages during each of the experimental visits in randomized order. Randomization will be completed using a research randomizer (randomizer.org), and the order that the drinks are consumed at each experimental visit will be different for each participant. Subjects will be blinded to which they are consuming. The investigators performing the tests will also be blinded to the order of test beverage administration. Subjects will be asked to maintain their dietary and lifestyle practices throughout the study, abstain from alcohol and recreational drugs throughout the study, and refrain from caffeine and stimulant usage except for that contained in the test beverages. More information regarding the test beverages are provided in the sub-section immediately below. In addition, a figure providing an overview of the study design/procedures has been included as an attachment.

At each experimental visit, subjects will come to the laboratory in a fasted state and provide a urine sample to validate their hydration status. Then, they will have their body composition assessed with a medical-grade bioelectrical impedance scale, complete questionnaires assessing their mood and energy, and then have their resting blood pressure and heart rhythm (using an electrocardiogram) assessed. Following these assessments, resting femoral artery blood flow will be evaluated using an ultrasound-based assessment in the thigh. Following this test, participants will consume a test beverage (e.g., the intervention) within 5 minutes. Following beverage consumption, they will complete assessments of maximal leg muscle static strength. They will then rest for approximately 30 minutes, and will have blood pressure, heart rate and rhythym (EKG), and blood flow evaluated again. After being instrumented with specialized sensors that measure muscle activity and heart rate, and a special mask that is used to capture the pulmonary gases that they expire for analyses, participants will complete a graded exercise test on a special exercise bike. The test will get progressively harder and proceed until they cannot continue exercise, and participants will wear the special sensors and mask for the entire duration of the test. They will also provide subjective assessments of their effort throughout the test. Immediately following completion of this test, they will again complete an assessment of their maximal leg muscle strength. Following a 5-minute rest period, they will complete a sustained, submaximal leg extension task for as long as possible at about 40% of their maximal effort. A blood pressure cuff on their arm will be used to measure blood pressure at the end of exercise. They will then complete one final maximal voluntary static strength assessment. After all exercise-related testing, a 15-minute observation period will immediately ensure. During this period, leg blood flow, resting blood pressure and heart rhythm (e.g., ECG), and assessments of mood, energy, and perceived exertion will be performed. Finally, 1-week nutrition, activity, and sleep logs, mood assessments, and instructions will be provided for them to complete during the week before they leave the laboratory.

Throughout the study, the study staff will contact participants via text or email with regular reminders regarding study procedures and their scheduled experimental visits. If they do not respond to reminders, study staff will follow-up with phone calls in order to ensure they are receiving the information provided and that they are still interested in participating.

Test Beverage Information The test beverages included in this study are commercially available beverages that are advertised to increase performance. These beverages include electrolyte enhanced water, and energy drinks that contain caffeine. These drinks are all commercially available, and will also include other ingredients including sugar/glucose, ginseng, guarana extract, L-carnitine, beta-alanine, L-citrulline, betaine, and B-vitamins. The subjects and the research staff administering the tests will be blinded to the drink that subjects are consuming. The total dose of caffeine in each test beverage will not exceed 200 mg. The specific beverages used in this study will include Monster Original Green Energy which contains 160 mg of caffeine, and Nutrabolt's Cellucor Carbonated C4 Energy which contains 200 mg of caffeine.

ELIGIBILITY:
Eligibility criteria (responses needed to be considered eligible in parentheses) are:

* Are you an assigned biological male? (Yes)
* Are you between the ages of 20 and 35 years? (Yes)
* Do you performed planned physical activity (i.e., planned walk/jog/run, bicycle ride, resistance exercise, sport participation, etc) on 3 or more days per week? (Yes)
* Do you consume 21 or more servings of >=6 fl ounces of caffeinated beverages each week? (No)
* Do you have a current illness that would impede participation in the study? (No)
* Has your doctor ever said that you have a heart condition or high blood pressure? (No)
* Do you feel pain in your chest at rest, during your activities of daily living, or when you do physical activity? (No)
* Do you lose balance because of dizziness (unrelated to over-breathing) or have you lost consciousness in the last 12 months (unrelated to a head injury)? (No)
* Do you currently have a bone, joint, or soft tissue injury that could be made worse by becoming more physically active? (No)
* Has your doctor ever said that you should only do physical activity if it is medically supervised? (No)
* Do you utilize nicotine or cannabis? (No)
* Do you currently use a prescription ADD/ADHD, anti-depressant, or other central acting medication, or were you previously diagnosed with ADD/ADHD, clinical depression, or other mental health condition? (No)
* Have you chronically (>6 months) abused illicit drugs or alcohol? (No)
* Are you currently being treated for metabolic syndrome or have you been clinically diagnosed with or taking medication for a metabolic-disorder including pre-diabetes, type II diabetes, high blood pressure, or obesity? (No)
* Have you been clinically diagnosed with a digestive disorder or sensitivity, or do you regularly utilize over-the-counter or dietary supplements to support gastrointestinal pain or discomfort? (No)
* Have you ever been diagnosed with an allergy to any ingredient present in the study treatments which are commercially available energy drinks, including but not limited to caffeine, artificial sweeteners (e.g., sucralose, acesulfame potassium), niacin, maltodextrin, ginseng? (No)
* Are you currently a competitive athlete? (No)
* Are you willing and unwilling and able to comply with the controls or experimental conditions of the study, as described in the informed consent document? (Yes)

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Maximal Exercise Performance | 50-minutes after the intervention
  Maximal oxygen consumption during ramp cycle test
Sub-maximal Exercise Performance | 50-minutes after the intervention
  Ventilatory Threshold during ramp cycle test
Fatiguing Isometric Exercise Performance | 65-minutes after the intervention
  Total impulse (Force*time) during sub-maximal isometric fatigue test at 40% of maximal force production

SECONDARY OUTCOMES:
Mood | 80-minutes after the intervention
  Total Mood Disturbance as Measured using the Profile of Mood States Short Form (POMS-SF)
Change in Systolic Blood Pressure | Pre-intervention, 40-minutes Post-intervention, 85-minutes Post-intervention
  Systolic Blood Pressure (mmHg)
Change in Diastolic Blood Pressure | Pre-intervention, 40-minutes Post-intervention, 85-minutes Post-intervention
  Diastolic Blood Pressure (mmHg)
Change in Heart Rate | Pre-intervention, 40-minutes Post-intervention, 85-minutes Post-intervention
  Heart Rate (bpm)
Change in Rate Pressure Product | Pre-intervention, 40-minutes Post-intervention, 85-minutes Post-intervention
  Rate Pressure Product (bpm*mmHg)
Change in QTc Interval | Pre-intervention, 40-minutes Post-intervention, 85-minutes Post-intervention
  QTc Interval measured by 12-lead ECG (ms)
Change in Leg Blood Flow | Pre-intervention, 40-minutes Post-intervention, and 75-minutes Post-Intervention
  mean femoral artery blood flow measured by high-resolution duplex ultrasonography

OTHER OUTCOMES:
Maximal Isometric Force Production | Pre-intervention, 65-minutes Post-Intervention, 70-minutes Post-Intervention, 74-minutes Post-Intervention
  Maximal Isometric Leg Extension Force Production
Time Completed During Fatiguing Isometric Exercise Performance | 72-min Post-intervention
  Time to Fatigue (s)
Force During Fatiguing Isometric Exercise Performance | 65-minutes after the intervention
  Average Submaximal Isometric Force (V)
Session Rating of Perceived Exertion | 80-minutes Post-intervention
  RPE across entire session as rated on scale of 0-10, with 10 representing maximal effort.
Adverse Events | 80-minutes Post-intervention
  Participants selected either "yes" or "no" to questions asking if they experienced any of the following: nausea, vomiting, headache, stomachache/bloating/gas, diarrhea, constipation, itching, fatigue, heart palpations, or other. If "yes" was selected, participants were then asked to mark how likely - possible, likely, or very likely - they believed that the adverse event/symptom was caused by the treatment beverage.
Blinding Efficacy | 80-minutes Post-intervention
  Participants were told that the three beverages they consumed were Monster Energy, C4 Energy, and Placebo, and were asked to indicate, to the best of their ability, in which visit they believed they had consumed each test beverage.
Change in Secondary ECG Characteristics | Pre-intervention, 40-minutes Post-intervention, 85-minutes Post-intervention
  PR and QRS interval (ms)

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Laboratory of Applied Physiology and Lifestyle Medicine, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data will be provided to other researchers upon reasonable request.

REFERENCES:
- [Background] https://www.nccih.nih.gov/health/energy-drinks
- [Background] Global energy drinks market: insights, market size, share, growth, trends analysis and forecast to 2021. AIM Market Insight. April 2015. Available at: https://www.researchandmarkets.com/research/mbbjvv/global_energy. Accessed December 20, 2017
- [Background] De Sanctis V, Soliman N, Soliman AT, Elsedfy H, Di Maio S, El Kholy M, Fiscina B. Caffeinated energy drink consumption among adolescents and potential health consequences associated with their use: a significant public health hazard. Acta Biomed. 2017 Aug 23;88(2):222-231. doi: 10.23750/abm.v88i2.6664. PMID 28845841
- [Background] Al-Shaar L, Vercammen K, Lu C, Richardson S, Tamez M, Mattei J. Health Effects and Public Health Concerns of Energy Drink Consumption in the United States: A Mini-Review. Front Public Health. 2017 Aug 31;5:225. doi: 10.3389/fpubh.2017.00225. eCollection 2017. PMID 28913331